CLINICAL TRIAL: NCT04579185
Title: Detailed Protocol: Evaluation of Transcranial Photobiomodulation for the Treatment of Pediatric Depression: An Open-Label Pilot Study
Brief Title: Transcranial Photobiomodulation for the Treatment of Pediatric Depression
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID, this study was not initiated
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Carrie Vaudreuil, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020P002694
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Depression
Keywords: light therapy; pediatric depression; depression; MDD
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcranial Photobiomodulation (Experimental): Transcranial Photobiomodulation--a noninvasive intervention in which near-infrared light (850 nanometer) is applied to forebrain.
  Interventions: Device: Transcranial Photobiomodulation

INTERVENTIONS:
Device: Transcranial Photobiomodulation — Transcranial Photobiomodulation--a noninvasive intervention in which near-infrared light (850 nanometer) is applied to forebrain.
  Other Names: Niraxx G1 Headband

SUMMARY:
An open label trial to assess the safety and efficacy of transcranial photobiomodulation (tPBM) in improving symptoms of depression in youth.

DETAILED DESCRIPTION:
Pediatric depression is a prevalent and morbid disorder estimated to affect up to 12% of youth in the United States by the time they reach adolescence. Recent research has documented that even minor symptoms of depression as captured through the Child Behavior Checklist (CBCL) Anxiety/Depression scale are strongly associated with the subsequent development of major depression. While treatments with antidepressants and psychotherapy are available, antidepressants can be associated with adverse effects including manic activation and psychosocial interventions are costly and not wide available. This state of affairs supports the search for safe and effective alternative treatments.

One such opportunity is transcranial LED therapy, also known as transcranial photobiomodulation (tPBM). The treatment consists of exposing the frontal brain to the tPBM bilaterally, which is hypothesized to enhance adenosine triphosphate (ATP) production in depressed subjects. tPBM is a non-ionizing electromagnetic wave. It is invisible, penetrates the skin and skull into brain tissue, is non-invasive, is minimally dissipated as thermal energy, and is mainly absorbed by specific chromophores. The benefits of tPBM are wavelength specific. A mitochondrial enzyme, the cytochrome c oxidase, is the primary chromophore for the tPBM, with a wavelength around 830 nm. The energy absorbed by the cytochrome c oxidase leads to increased ATP production through the respiratory chain. Ultimately, the increased ATP is thought to lead to increased energy metabolism for the cell, and it is hypothesized that a signaling cascade is activated promoting cellular plasticity and cytoprotection. These properties of the tPBM have led to novel therapeutic applications in psychiatry. A preliminary open label study in 10 depressed subjects has shown that the tPBM was safe, effective and well tolerated in depressed adults. Further research confirmed these findings and shown tPBM therapy to be a promising intervention for adults with MDD. However, whether this non-invasive intervention may be safe and effective in pediatric depression remains unknown.

To this end the investigators propose a pilot study is to evaluate whether tPBM is safe and effective in the treatment of pediatric depression. This study will enroll 30 youth of both sexes 6-17 years with active symptoms of depression as assessed through elevated scores on the CBCL Anxiety/depression scale. Based on the adult literature, investigators hypothesize that it will be safe and effective in this population.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children aged 6- 17 years
* A CBCL T score of ≥ 60 on the Anxious/Depressed scale
* Current treatment with a psychotropic medication or psychological treatment will be allowed provided that no medication or psychological treatment changes occur during the study

Exclusion Criteria:

* Clinically unstable current psychiatric conditions judged to be a serious safety risk to self or others such as active suicidal ideation, psychosis or mania
* Subjects with an unstable medical condition that requires clinical attention
* The subject has a significant skin condition at the procedure sites (i.e., hemangioma, scleroderma, psoriasis, rash, open wound or tattoo).
* Inadequate command of the English language
* History of neurological injury or disease
* Impaired intellectual capacity (clinically determined)
* The subject has an implant of any kind in the head (e.g. stent, clipped aneurysm, embolised AVM, implantable shunt - Hakim valve).
* Any use of light-activated drugs (photodynamic therapy) within 14 days prior to study enrollment (in US: Visudine (verteporfin) - for age related macular degeneration; Aminolevulinic Acid- for actinic keratoses; Photofrin (porfimer sodium) - for esophageal cancer, non-small cell lung cancer; Levulan Kerastick (aminolevulinic acid HCl) - for actinic keratosis; 5-aminolevulinic acid (ALA)- for non-melanoma skin cancer
* Investigator and his/her immediate family, defined as the investigator's spouse, parent, child, grandparent, or grandchild

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Efficacy-Major Depressive Disorder (Clinical Global Impression - Major Depressive Disorder) | Baseline to Week 8
  To evaluate the efficacy of transcranial photobiomodulation in treatment of depression. The Clinical Global Impression Scale rates symptoms of depression from a scale of 1 (normal, not at all ill) to 7 (among the most extremely ill patients), with higher scores on this scale indicating a worse outcome.

SECONDARY OUTCOMES:
Safety (The Transcranial Photobiomodulation Self-Report Questionnaire) | Baseline to Week 8
  To assess the safety of transcranial photobiomodulation for treatment of depression. The Transcranial Photobiomodulation (tPBM) Self-Report Questionnaire rates the patient's comfort/discomfort with the tPBM on a scale of 0 (not discomfort) to 5 (extreme discomfort), with higher scores on this scale indicating a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Vaudreuil, MD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barrett B, Byford S, Knapp M. Evidence of cost-effective treatments for depression: a systematic review. J Affect Disord. 2005 Jan;84(1):1-13. doi: 10.1016/j.jad.2004.10.003. PMID 15620380
- [Background] Cassano P, Petrie SR, Hamblin MR, Henderson TA, Iosifescu DV. Review of transcranial photobiomodulation for major depressive disorder: targeting brain metabolism, inflammation, oxidative stress, and neurogenesis. Neurophotonics. 2016 Jul;3(3):031404. doi: 10.1117/1.NPh.3.3.031404. Epub 2016 Mar 4. PMID 26989758
- [Background] Eells JT, Henry MM, Summerfelt P, Wong-Riley MT, Buchmann EV, Kane M, Whelan NT, Whelan HT. Therapeutic photobiomodulation for methanol-induced retinal toxicity. Proc Natl Acad Sci U S A. 2003 Mar 18;100(6):3439-44. doi: 10.1073/pnas.0534746100. Epub 2003 Mar 7. PMID 12626762
- [Background] Frye MA, Helleman G, McElroy SL, Altshuler LL, Black DO, Keck PE Jr, Nolen WA, Kupka R, Leverich GS, Grunze H, Mintz J, Post RM, Suppes T. Correlates of treatment-emergent mania associated with antidepressant treatment in bipolar depression. Am J Psychiatry. 2009 Feb;166(2):164-72. doi: 10.1176/appi.ajp.2008.08030322. Epub 2008 Nov 17. PMID 19015231
- [Background] Leverich GS, Altshuler LL, Frye MA, Suppes T, McElroy SL, Keck PE Jr, Kupka RW, Denicoff KD, Nolen WA, Grunze H, Martinez MI, Post RM. Risk of switch in mood polarity to hypomania or mania in patients with bipolar depression during acute and continuation trials of venlafaxine, sertraline, and bupropion as adjuncts to mood stabilizers. Am J Psychiatry. 2006 Feb;163(2):232-9. doi: 10.1176/appi.ajp.163.2.232. PMID 16449476
- [Background] Merikangas KR, He JP, Burstein M, Swanson SA, Avenevoli S, Cui L, Benjet C, Georgiades K, Swendsen J. Lifetime prevalence of mental disorders in U.S. adolescents: results from the National Comorbidity Survey Replication--Adolescent Supplement (NCS-A). J Am Acad Child Adolesc Psychiatry. 2010 Oct;49(10):980-9. doi: 10.1016/j.jaac.2010.05.017. Epub 2010 Jul 31. PMID 20855043
- [Background] Mochizuki-Oda N, Kataoka Y, Cui Y, Yamada H, Heya M, Awazu K. Effects of near-infra-red laser irradiation on adenosine triphosphate and adenosine diphosphate contents of rat brain tissue. Neurosci Lett. 2002 May 3;323(3):207-10. doi: 10.1016/s0304-3940(02)00159-3. PMID 11959421
- [Background] Schiffer F, Johnston AL, Ravichandran C, Polcari A, Teicher MH, Webb RH, Hamblin MR. Psychological benefits 2 and 4 weeks after a single treatment with near infrared light to the forehead: a pilot study of 10 patients with major depression and anxiety. Behav Brain Funct. 2009 Dec 8;5:46. doi: 10.1186/1744-9081-5-46. PMID 19995444
- [Background] Uchida M, Fitzgerald M, Woodworth H, Carrellas N, Kelberman C, Biederman J. Subsyndromal Manifestations of Depression in Children Predict the Development of Major Depression. J Pediatr. 2018 Oct;201:252-258.e1. doi: 10.1016/j.jpeds.2018.05.049. Epub 2018 Jul 13. PMID 30007773
- [Background] Zhang Q, Ma H, Nioka S, Chance B. Study of near infrared technology for intracranial hematoma detection. J Biomed Opt. 2000 Apr;5(2):206-13. doi: 10.1117/1.429988. PMID 10938785